CLINICAL TRIAL: NCT00970437
Title: A Comparison of Cognitive Behavioral Analysis System of Psychotherapy (CBASP) and System of Supportive Psychotherapy (SYSP) for Early Onset Chronic Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Elisabeth Schramm, PhD, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKF001906
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Chronic Major Depressive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBASP (Active Comparator): CBASP as the experimental intervention will follow a manual (McCullough, 2000; German version: Schramm et al., 2006). The approach is specifically tailored for the treatment of chronic forms of depression, particularly with early-onset by focusing on the problems resulting from an inhibition of maturation in early childhood and by using the therapeutic relationship in a personal, disciplined way as well as other specific techniques (e.g. Interpersonal Discrimination Exercise, Situation Analysis). CBASP integrates behavioural, cognitive, and interpersonal strategies.
  Interventions: Behavioral: Cognitive Behavioral Analysis System of Psychotherapy
- SYSP (Placebo Comparator): The comparator for CBASP is SYSP, a system of supportive psychotherapy, an active but less specific, manualized control treatment. SYSP - defined as non-interpersonal and non-cognitive-behavioral therapy - resembles supportive clinical management, client-centered therapy, counseling, and psychoeducation about depression. There is no specific explanatory mechanism for treatment effect offered to the patient and it does not focus on specific themes.
  Interventions: Behavioral: System of Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Analysis System of Psychotherapy — Duration of intervention per patient: 20 weeks acute treatment (n=24 sessions) followed by 28 weeks of continuation treatment (n=8 sessions) Follow-up per patient: 48 weeks after randomisation
  Arms: CBASP
Behavioral: System of Supportive Psychotherapy — Duration of intervention per patient: 20 weeks acute treatment (n=24 sessions) followed by 28 weeks of continuation treatment (n=8 sessions) Follow-up per patient: 48 weeks after randomisation
  Other Names: Brief Supportive Psychotherapy
  Arms: SYSP

SUMMARY:
The purpose of this study is to compare the efficacy of the Cognitive Behavioural Analysis System of Psychotherapy (CBASP) with the non-specific System of Supportive Psychotherapy (SYSP)in early onset chronically depressives.

DETAILED DESCRIPTION:
Effective treatment strategies for chronic depression are urgently needed since it is not only a common and particularly disabling disorder, but is also considered treatment resistant by most clinicians. There are only a few studies on chronic depression indicating that traditional interventions are not as effective as in acute, episodic depression. In addition, most of the studies had methodological weaknesses, such as the very short courses of psychotherapy. Usually, chronic depression begins early in life, is often associated with early interpersonal trauma, and results in an even more substantial human capital loss than the late-onset group. Furthermore, it shows a weak response to medication and a high rate of relapse after an initial response. With the present multicentre study, the efficacy of the only specific psychotherapy for chronic depression (Cognitive Behavioural Analysis System of Psychotherapy/CBASP) is compared with a non-specific System of Supportive Psychotherapy/SYSP in early onset chronically depressives. CBASP faired very well in one large trial but has never been directly compared to a non-specific psychotherapeutic control. Another innovative aspect of the study is the use of an extended course of psychotherapy (32 sessions). Primary hypothesis: CBASP is more effective in reducing depressive symptoms than SYSP.

A naturalistic study following up the patients of the trial up to two years after termination of the study treatments is performed in order to investigate the long-term effectiveness of CBASP compared to the System of Supportive Psychotherapy. The primary outcome of this follow-up study is the rate of well-weeks (weeks with no or minimal depression symptoms) during the two years after termination of the study treatments as measured with the Longitudinal Interval Follow-up Evaluation (LIFE) Interview

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV criteria for a current episode of chronic MDD, MDD superimposed on a pre-existing dysthymic disorder or recurrent MDD with incomplete remission between episodes in a patient with a current MDD and a total duration of at least 2 years.
2. Early onset of the disorder according to DSM-IV (onset before the age of 21)
3. Age between 18 and 65
4. A score of at least 20 on the 24-item HRSD at screening and, after a 2-week drug-free period, at baseline
5. Fluent in German language
6. Provide informed consent

Exclusion Criteria:

1. Acute risk for suicide (as opposed to suicidal thoughts) assessed according to clinical practice guidelines. Suicidal patients are eligible, as long as outpatient treatment is deemed safe by the clinician.
2. A history of psychotic symptoms, bipolar disorder, or organic brain disorders
3. A primary diagnosis of another axis I disorder including anxiety disorders (e.g. Posttraumatic Stress Disorder), or any severe substance-related abuse or dependence disorder as evaluated with the SCID-I
4. Antisocial, schizotypical, or borderline personality disorder (SCID-II);
5. Severe cognitive impairment
6. Absence of a response to previous adequate trial of CBASP, and/or SYSP
7. Other ongoing psychotherapy or medication
8. A serious medical condition (i.e. a history of seizures, severe head trauma, stroke or heart attack within six months before the study began)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2010-04; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms as measured by the HRSD (24-item Hamilton Rating Scale of Depression) | 20 weeks after randomization (after acute treatment phase)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Schramm, PhD, Principal Investigator — University Medical Center Freiburg, Department of Psychiatry and Psychotherapy; Martin Härter, MD, PhD, Principal Investigator — University Medical Center Hamburg
Locations (1):
- University Medical Center Freiburg, Department of Psychiatry and Psychotherapy, Freiburg im Breisgau, Germany

REFERENCES:
- [Result] Schramm E, Kriston L, Zobel I, Bailer J, Wambach K, Backenstrass M, Klein JP, Schoepf D, Schnell K, Gumz A, Bausch P, Fangmeier T, Meister R, Berger M, Hautzinger M, Harter M. Effect of Disorder-Specific vs Nonspecific Psychotherapy for Chronic Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Mar 1;74(3):233-242. doi: 10.1001/jamapsychiatry.2016.3880. PMID 28146251
- [Derived] Echterhoff J, Kriston L, Klein JP, Harter M, Schramm E, Schumacher L. Symptom-specific improvement across therapies and their putative mediators: A mediation network intervention analysis. Psychother Res. 2025 Apr;35(4):546-557. doi: 10.1080/10503307.2024.2320349. Epub 2024 Mar 3. PMID 38431848
- [Derived] Schumacher L, Klein JP, Elsaesser M, Harter M, Hautzinger M, Schramm E, Kriston L. Implications of the Network Theory for the Treatment of Mental Disorders: A Secondary Analysis of a Randomized Clinical Trial. JAMA Psychiatry. 2023 Nov 1;80(11):1160-1168. doi: 10.1001/jamapsychiatry.2023.2823. PMID 37610747
- [Derived] Humer E, Schramm E, Klein JP, Harter M, Hautzinger M, Pieh C, Probst T. Effects of alliance ruptures and repairs on outcomes. Psychother Res. 2021 Nov;31(8):977-987. doi: 10.1080/10503307.2021.1874070. Epub 2021 Jan 17. PMID 33455531
- [Derived] Meister R, Lanio J, Fangmeier T, Harter M, Schramm E, Zobel I, Hautzinger M, Nestoriuc Y, Kriston L. Adverse events during a disorder-specific psychotherapy compared to a nonspecific psychotherapy in patients with chronic depression. J Clin Psychol. 2020 Jan;76(1):7-19. doi: 10.1002/jclp.22869. Epub 2019 Oct 1. PMID 31576565
- [Derived] Assmann N, Schramm E, Kriston L, Hautzinger M, Harter M, Schweiger U, Klein JP. Moderating effect of comorbid anxiety disorders on treatment outcome in a randomized controlled psychotherapy trial in early-onset persistently depressed outpatients. Depress Anxiety. 2018 Oct;35(10):1001-1008. doi: 10.1002/da.22839. Epub 2018 Sep 10. PMID 30199128
- [Derived] Eich HS, Kriston L, Schramm E, Bailer J. The German version of the helping alliance questionnaire: psychometric properties in patients with persistent depressive disorder. BMC Psychiatry. 2018 Apr 23;18(1):107. doi: 10.1186/s12888-018-1697-8. PMID 29685124
- [Derived] Erkens N, Schramm E, Kriston L, Hautzinger M, Harter M, Schweiger U, Klein JP. Association of comorbid personality disorders with clinical characteristics and outcome in a randomized controlled trial comparing two psychotherapies for early-onset persistent depressive disorder. J Affect Disord. 2018 Mar 15;229:262-268. doi: 10.1016/j.jad.2017.12.091. Epub 2018 Jan 4. PMID 29329058
- [Derived] Schramm E, Hautzinger M, Zobel I, Kriston L, Berger M, Harter M. Comparative efficacy of the Cognitive Behavioral Analysis System of Psychotherapy versus supportive psychotherapy for early onset chronic depression: design and rationale of a multisite randomized controlled trial. BMC Psychiatry. 2011 Aug 17;11:134. doi: 10.1186/1471-244X-11-134. PMID 21849054